CLINICAL TRIAL: NCT04062721
Title: Feasibility and Safety of Local Immunomodulation Combined With Radiofrequency Ablation for Unresectable Colorectal Liver Metastases: A Monocentric Phase I Trial
Brief Title: Local Immunomodulation After Radiofrequency of Unresectable Colorectal Liver Metastases
Acronym: LICoRN-01
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19RME-LICORN
Record Dates: First submitted 2019-06-18; First posted 2019-08-20 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Unresectable Colorectal Liver Metastases
Keywords: Colorectal cancer; Liver metastases; Radiofrequency; Immunomodulation
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Drug Therapy; Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chemotherapy + RFA + in situ immunotherapy (Experimental): Patients with non-resectable CRC liver-only metastases.
  Interventions: Drug: Chemotherapy; Procedure: Radiofrequency ablation (RFA); Drug: In situ immunotherapy

INTERVENTIONS:
Drug: Chemotherapy — Chemotherapy (at the investigator's choice) for ≥ 2 months before RFA (with controlled disease) and resumed 4-6 weeks after RFA to achieve 6-month total duration.
Procedure: Radiofrequency ablation (RFA) — Complete macroscopic ablation by RFA.
Drug: In situ immunotherapy — Hydrogel combining TLR or NOD2 agonist and GM-CSF will be injected in 1, 2 or 3 distinct lesions after RFA.

SUMMARY:
The main objective of this trial is to determine feasibility and tolerance of the human body to RFA associated with local immunomodulation carried out using a thermoreversible hydrogel combined with 2 immunomodulators, GMCSF and Mifamurtide.

The main endpoint of the study is the feasibility, the frequency and the nature of per and post-operative adverse events of the in situ injection of an immunomodulatory hydrogel after radiofrequency of unresectable colorectal liver metastases.

The secondary objective is one-year progression free survival rate.

DETAILED DESCRIPTION:
Early clinical trials of immunotherapy in colorectal cancer (CRC) have provided first evidence of activity of adoptive cell vaccines combining inactivated autologous tumor cells and BCG, a Toll Like Receptor (TLR) agonist. RFA induces tumor cell necrosis and apoptosis, leading to the activation of anti-tumoral immunity through the release, exposure or denaturation of tumor antigens, which are captured by dendritic cells. Associated pro-inflammatory effects increase the anti-tumoral immune response but remain insufficient to avoid recurrence. In a preclinical study in an aggressive rectal cancer model, complete and long-lasting tumor responses were achieved after RFA combined with in situ injection of an immunomodulatory hydrogel combining a TLR agonist and GM-CSF. These results were obtained without further adjuvant therapy after complete clearance of macroscopic liver lesions by RFA(1,2). BCG, bacteria Protein Derivatives can be used as TLR or NOD2 agonists. The hypothesis of the study is that local immunotherapy may reduce recurrence rates after RFA in patients with unresectable liver metastases from CRC.

Thermal ablation by RFA may be used as an inducer of anti-tumor immune response and the combination with immunomodulators such as a TLR or NOD2 agonists and GM-CSF may improve its efficacy. In the recent preclinical study, the efficacy has been demonstrated on distant lesions (so-called abscopal effect) of two immunomodulators combined in a muco-adherent hydrogel, injected in a RFA-treated tumor. The treatment was safe. Complete macroscopic ablation by RFA combined with in situ immunomodulators may be able to prime an effective immune response capable of eradicating the microscopic residual disease.

This study is an open label, quasi-experimental, non-randomized, single-arm trial.

Will be included patients with unresectable colorectal hepatic metastases, without extra hepatic localization. A complete clearance of lesions must be obtained by the use of radiofrequency alone or combined with surgery.

These patients will have complete destruction, by laparotomy, by radiofrequency alone or associated with surgery of all the liver metastases detectable at the time of treatment.

12 patients meeting inclusion criteria and not exclusion ones will be included and expected to be valuable patients. 3 subgroups of 4 patients each will receive an immunogel injection in 1, 2 and 3 metastases respectively as dose escalation. The primary endpoints will be collected in post-operative course until 3 months however, the patients will be followed in the trial until 12 months after RFA.

The radiofrequency of one, two or three lesions (dose escalation) selected on preoperative imaging, will be followed by injection, under ultrasound control via a coaxial device, of 5 ml (lesion < 2 cm) or 10 ml (lesion ≥ 2 cm) of thermoreversible gel vectorising 2 immunomodulators, mifamurtide (8 µg / ml) and GMCSF (25 µg / ml). The choice of mifamurtide, the liposomal form of the smallest synthetic immunogenic derivative of the wall of mycobacteria, is justified by the need to replace BCG, used in preclinical studies, by an inert immunomodulator. This compound has demonstrated its clinical efficacy in anti-tumor immunotherapy. GMCSF was largely used in antitumor immunotherapies studies and platforms.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained from the patient prior to performing any protocol-related procedures, including screening evaluations;
2. Willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up;
3. Histologically or cytologically proven CRC;
4. Non-resectable liver metastases from CRC without detectable extra-hepatic disease, on abdomino-pelvic computed tomography (CT) or magnetic resonance imaging (MRI) and chest CT by the consulting hepatobiliary surgeon and radiologist. Unresectability is defined as no possibility to completely resect all tumor lesions;
5. Age ≥ 18 years;
6. ECOG PS 0-1;
7. Controlled disease (stability or objective response) with chemotherapy (≥ 2 months) for liver metastases;
8. Liver metastases ≥ 3 and <10, including ≥ 3 lesions accessible to RFA;
9. Maximum diameter of 4 cm for lesions to be treated by RFA;
10. Metastatic involvement of the liver ≤50%;
11. Complete treatment of all liver lesions judged possible, either by RFA alone or by combination with resection of resectable lesions and RFA of the remaining non-resectable liver deposits;
12. Measurable or evaluable (radiologically detectable disease which does not fulfill RECIST criteria for measurable disease) lesions according to RECIST v1.1 criteria (CT-scan < 4 weeks);
13. Adequate organ function, as defined by the following:

    1. Serum aspartate aminotransferase (AST) and serum alanine aminotransferase (ALT) < 3 x upper limit of normal (ULN);
    2. Total serum bilirubin < 1.5 ULN;
    3. Prothrombin ratio > 70%;
    4. Serum albumin ≥ 30 g/L;
    5. Hemoglobin ≥ 10.0 g/dl;
    6. White blood cell count (WBC) ≥ 3,000/μL;
    7. Absolute neutrophil count (ANC) ≥ 1,500/μL;
    8. Platelets ≥ 150,000/μL;
    9. Serum creatinine ≤ 1.5 ULN or creatinine clearance > 50 mL/min (MDRD);
14. Any other prior therapy directed at the malignant tumor, including chemotherapy; chemoembolization therapy, molecular targeted therapy (including antiangiogenics), and radiotherapy, must be discontinued at least 2 weeks prior to registration and at least 3 weeks before day 1 on trial;
15. Life expectancy ≥ 3 months;
16. Evidence of post-menopausal status, negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause;
17. Women participants of childbearing potential must have a negative serum pregnancy test within the 7 days prior to the first treatment administration;
18. Registration in a national health care system.

Exclusion Criteria:

1. Any other malignancy in the past 10 years (except carcinoma of the cervix in situ or no melanoma skin cancer);
2. Clinical significant cardiovascular disease;
3. Uncontrolled hypertension, bleeding disorders or coagulopathy, active infection;
4. Major surgical procedures within 28 days before RFA;
5. Concurrent enrolment in another clinical study, unless it is an observational (noninterventional) or supportive care clinical study or during the follow-up period of an interventional study;
6. Receipt of the last dose of anticancer therapy (investigational product, chemotherapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies) ≤ 21 days prior to the RFA. If sufficient wash-out time has not occurred due to the schedule or pharmacokinetics properties of an agent, a longer wash-out period will be required;
7. Histology other than adenocarcinoma;
8. Extensive tumor massively replacing both entire lobes;
9. Obstructive jaundice (bilirubin > 1.5 ULN) without adequate biliary drainage;
10. Any unresolved toxicity NCI CTCAE Grade ≥ 2 from previous anticancer therapy with the exception of alopecia, neuropathy, and the laboratory values defined in the inclusion criteria;
11. History of allogenic organ transplantation;
12. Any systemic steroid therapy whatever the duration of this corticotherapy;

    Note: The following are exceptions to this criterion:
    * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
    * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication);
13. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies); Note: Patients with past HBV infection or resolved HBV infection (defined as having a negative HBsAg test and a positive hepatitis B core antigen [HBc] antibody test) are eligible.

    Note: Patients positive for HCV antibody are eligible only if polymerase chain reaction testing is negative for HCV ribonucleic acid (RNA).
14. Diagnosis of any second malignancy within the last 5 years, except for adequately treated basal cell or squamous cell skin cancer, or in situ carcinoma of the cervix uteri;
15. Known active central nervous system metastases and/or carcinomatous meningitis; patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least 4 weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids > 10 mg/day of prednisone or equivalent for at least 14 days prior to trial treatment;
16. Uncontrolled massive pleural effusion or massive ascites;
17. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]), that has required systemic treatment (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs); Note: Patients with vitiligo, alopecia, or any chronic skin condition that does not require systemic therapy are exception to this criterion.

    History of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone may be eligible. Controlled Type 1 diabetes mellitus on a stable insulin regimen may be eligible.
18. Uncontrolled undercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent;
19. Live vaccine administration, excepted BCG, within 30 days prior to the RFA;
20. Known or suspected allergy or hypersensitivity to any of the study component or any of the study vaccine excipients;
21. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with participation for the full duration of the trial, or is not in the best interest of the participant, in the opinion of the treating investigator;
22. Pregnancy/lactation;
23. Tutelage or guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | at 3 months
  All grade and severe (grade 3-5) toxicities, according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0 including post-operative and immune-related complications within 3 months after surgery.

SECONDARY OUTCOMES:
Progression free survivor (PFS) rate at 12 months | at 12 months
  Progression free survivor (PFS) rate at 12 months assessed by centralized review of computed tomography (CT)-scan imaging in evaluable patients. Evaluable patients to determine PFS at 12 months will be:
  * Patients alive at 12 months and with a documented progression on CT-scan available at 12 months or before;
  * Patients alive at 12 months and without a documented progression on CT-scan available at 12 months;
  * Patients dead within 12 months.
  * The PFS rate at 12 months will be defined as the proportion of patients who will be alive and without disease progression at 12 months after RFA, according to RECIST v1.1, assessed by centralized review of CT-scan imaging.
Median PFS | at 12 months
  Time from the date of RFA to progression according to RECIST v1.1, assessed by centralized review of CT-scan imaging, or death for any reason, whichever occurs first.
Median overall survival (OS) | at 24 month
  Time from the date of RFA to date of death.
Response rate | at 12 months and 24 months
  According to RECIST v1.1.
Potential predictive biomarkers | at baseline and every two months until 24 months
  Will be collected at baseline and every two months until 24 months after the day of RFA, biological data (blood and tumor tissue) for tumorous markers.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Malafosse, MD, Principal Investigator — Digestive Surgery Department, Ambroise Pare University Hospital, Boulogne-Billancourt, France; Cindy NEUZILLET, MD, PhD, Study Director — Digestive Surgery Department, Ambroise Pare University Hospital, Boulogne-Billancourt, France
Locations (1):
- Digestive Surgery Department, Ambroise Pare University Hospital, APHP, Boulogne-Billancourt, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lemdani K, Seguin J, Lesieur C, Al Sabbagh C, Doan BT, Richard C, Capron C, Malafosse R, Boudy V, Mignet N. Mucoadhesive thermosensitive hydrogel for the intra-tumoral delivery of immunomodulatory agents, in vivo evidence of adhesion by means of non-invasive imaging techniques. Int J Pharm. 2019 Aug 15;567:118421. doi: 10.1016/j.ijpharm.2019.06.012. Epub 2019 Jun 6. PMID 31176849
- [Background] Lemdani K, Mignet N, Boudy V, Seguin J, Oujagir E, Bawa O, Peschaud F, Emile JF, Capron C, Malafosse R. Local immunomodulation combined to radiofrequency ablation results in a complete cure of local and distant colorectal carcinoma. Oncoimmunology. 2019 Jan 10;8(3):1550342. doi: 10.1080/2162402X.2018.1550342. eCollection 2019. PMID 30723580